CLINICAL TRIAL: NCT03107429
Title: A Pilot Crossover Study in Healthy Volunteers to Assess the Effect of Acetazolamide on Intraocular Pressure After Being in the Trendelenburg Position.
Brief Title: Effect of Acetazolamide on Intraocular Pressure After Being in the Trendelenburg Position.
Acronym: TaPPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: C12022015 SoM NDDC TaPPs
Record Dates: First submitted 2017-02-21; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: IOP
Keywords: Trendelenburg; Laparoscopic colorectal surgery; POVL
MeSH Terms: interventions — Acetazolamide; Head-Down Tilt

STUDY DESIGN:
Intervention Model Description: A pilot blinded randomised cross-over study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo and Acetazolamide tablets were placed into capsules that were the same by the Pharmacy department. A separate investigator generated a randomisation list for 11 volunteers to decide if a placebo or acetazolamide will be taken on Day 1. They then created envelopes with the corresponding medication in Day 1 and the other in Day 2 and these were marked as Volunteer 1, 2, 3 etc. The randomisation list was sealed and kept with each investigator so they could be accessed if required due to any adverse events.
  The volunteers will be recruited and both the investigators and the volunteers were blinded to what was received on each study day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo and Trendelenburg Position (Active Comparator): Volunteers received placebo medication and placed in Trendelenburg.
  IOP will be measured. Participants will then be administered with a placebo and after 2.5 hours will be placed in 17 degrees head-down position for a minimum of 1 hour and maximum 4 hours. Repeat IOP measure will be taken whilst still in the Trendelenburg position after 5 mins and then every 30 minutes.
  Interventions: Drug: Placebo; Other: Trendelenburg Position
- Acetazolamide and Trendelenburg Position (Experimental): Volunteer given acetazolomide and placed in Trendelenburg position and IOP measured.
  IOP will be measured. Participants will then be administered with acetazolamide and after 2.5 hours placed in 17 degrees head-down position for a minimum of 1 hour and maximum 4 hours. Repeat IOP measure will be taken whilst still in the Trendelenburg position after 5 mins and then every 30 minutes.
  Interventions: Drug: Acetazolamide; Other: Trendelenburg Position

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide tablets were placed in capsules to make them look similar to placebo.
  Other Names: Diamox
  Arms: Acetazolamide and Trendelenburg Position
Drug: Placebo — Placebo was a sugar based placebo placed in a capsule.
  Other Names: Placebo arm, Placebo and Trendelenburg.
  Arms: Placebo and Trendelenburg Position
Other: Trendelenburg Position — Placed in Trendelenburg Position

SUMMARY:
Perioperative vision loss following laparoscopic colorectal surgery is rare but has been reported. Studies show Trendelenburg positioning during surgery can produce a significant rise in the IOP, and this rise is thought to be a possible factor. Acetazolamide decreases IOP by reducing the formation of aqueous humour.

Aims:

To investigate if acetazolamide reduces the IOP rise resulting from Trendelenburg positioning.

Methods:

A randomised cross-over blinded pilot study. Nine healthy volunteers were randomised to start with the placebo or Acetazolamide with a 5 days' washout period. Baseline IOP was measured on both days. After 1.5 hours of taking the medication, volunteers lay head-down at 17 degrees' for 4 hours and IOP measurements repeated. This reading was subtracted from the baseline to give a 'change in IOP'.

DETAILED DESCRIPTION:
Background:

Laparoscopic (keyhole) bowel surgery often requires positioning patients on the operating table in very steeply angled positions for up to four or more hours. There have been case reports of patients suffering cognitive impairment after surgery with long periods of Trendelenburg (person is lying flat at an incline where their head lies lower than their feet) positioning.

Evidence from other fields of surgery suggests that "head-down" positions can produce a significant rise in the intraocular pressure. Transient vision problems and loss of sight has been reported following surgery is rare instances, including one case after laparoscopic colorectal resection. The cause of this is not fully understood, but rises in intraocular pressure (IOP) has been suggested as a possible factor. This may be particularly relevant in patients who have pre-existing high baseline IOP as a result of glaucoma. Studies looking at the effect of Trendelenburg positioning have shown that there is an increase in IOP. This study is to assess the effect of acetazolamide on the IOP rise after being placed in the Trendelenburg position. Acetazolamide is a carbonic anhydrase inhibitor which is used to treat glaucoma. The drug works by decreasing aqueous humour formation. It can be given as eye drops (but the absorption of this is variable and therefore so is the effect), orally and intravenously. The oral dose can be given as a one off dose or a divided dose. Maximum onset of IOP reduction occurs 2 to 5 hours after taking an oral dose and duration is 6-8 hours.

Aims:

This study aims to investigate the effect of acetazolamide on the IOP rise whilst in the Trendelenburg position.

Experimental protocol and methods:

This will be a pilot randomised crossover study with 9 healthy volunteers recruited and randomised to either Group 1 or Group 2. Group 1 will start with the Control Day; Group 2 will start with the Intervention Day. On the Control Day, a baseline IOP using a Tonopen XL will be taken. They will then be placed in 17 degrees head-down position 2.5hours after a placebo is administered for a minimum of 1 hour and a maximum of 4 hours. Repeat IOP measure will be taken whilst in the Trendelenburg position after 5 minutes, and then every 30 minutes from the start of Trendelenburg position. On the Intervention Day, baseline IOP will be taken, they will then be 500mgs of acetazolamide. After 2.5 hours, the volunteers will then be placed in the Trendelenburg position at 17 degrees for position for a minimum of 1hour and a maximum of 4 hours. Repeat IOP measure will be taken whilst in the Trendelenburg position after 5 minutes, and then every 30 minutes from the start of Trendelenburg position.

Inclusion criteria:

Healthy volunteers, aged 18 and over

Exclusions criteria

Pregnancy Breast Feeding Hepatic impairment Patients with pre-existing conditions affecting IOP regulation eg Glaucoma, previous eye surgery Regular medication affecting IOP Under the age of 18 Refusal to give written informed consent

Measurable endpoints/ statistical power

Primary endpoint: Comparison of IOP pressure before and after being placed in the Trendelenburg position between the two days - Day 1 volunteers will be administered with a placebo before being placed in the Trendelenburg position and Day 2 after acetazolamide has been administered.

Power: Bucci et al compared the effect of oral acetazolamide on IOP on 22 patients. They detected a 3.7mmHg decrease in IOP after 2 hours. Using this study, we powered our study to require 18 patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 and over

Exclusion Criteria:

* Pregnancy
* Breast Feeding
* Hepatic impairment
* Patients with pre-existing conditions affecting IOP regulation eg Glaucoma, previous eye surgery
* Regular medication affecting IOP
* Under the age of 18
* Refusal to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of IOP pressure during Trendelenburg position after placebo and acetazolamide at each given time point outlined in methods. | 6 days. 2 Days involved in study (6 hours each) and a minimum of 5 days between study days to allow 'wash-out period' of drug.
  IOP measurements will be taken at each described time point on both study days and the difference in IOP measurement after acetazolamide will be compared to those after placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Parveen Vitish-Sharma, MRCS MSc, Principal Investigator — NDDC BRU

IPD SHARING:
Plan to Share IPD: No